CLINICAL TRIAL: NCT03388099
Title: Impact of Gonadotrophin REceptor Polimorphisms on the Relationship Between Serum AMH and Ovarian Response
Acronym: GREPAMOR
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1706-VLC-058-EB
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: antimüllerian Hormone and Gonadotrophin Receptor Polymorphism as Predictors of Ovarian Response
Keywords: gonadotrophin receptor polymorphism; antimüllerian hormone; ovarian response; ovarian stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with FSH/LH polymorphisms: Infertile patients will undergo an ovarian stimulation with FSH and/or hMG. Doses will be chosen according to BMI, Antral follicle count, AMH and age.
- patients without FSH/LH polymorphisms: Infertile patients will undergo an ovarian stimulation with FSH and/or hMG. Doses will be chosen according to BMI, Antral follicle count, AMH and age.

SUMMARY:
Aim of study: To compare the relationship between serum AMH and ovarian response for IVF with the GnRH antagonist protocol in patients who are carriers of FSH and/or LH receptor polymorphisms with those that are not.

DETAILED DESCRIPTION:
Serum AMH has shown to have a high predictive capability of the ovarian response to stimulation for IVF. On the other hand, patients who are carriers of polymorphisms in the FSH and LH receptors, have shown to need higher doses of gonadotrophins for ovarian stimulation. The proportion of carriers has been described to be around 20% of the population. Nevertheless, the determination of these polymorphisms is not performed in routine practice. It is unknown if their presence affects to the relationship between serum AMH levels and ovarian response.

This is a prospective, single center, non-interventional, cohorts study.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age presenting to IVF clinic
* BMI of 18-35 kg/m2
* Having been tested for serum AMH with the Elecsys assay
* Being planned to undergo ovarian stimulation cycle for IVF with the GnRH antagonist protocol
* Signed written informed consent or waiver

Exclusion Criteria:

* Current or past disease affecting ovaries, gonadotropin or sex steroid
* Current hormone therapy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women will undergo an ovarian stimulation for IVF treatment
Study Population: Infertile Patients undergoing IVF treatments
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Gonadotrophin receptor polymorphisms and ovarian response and AMH value | 1 year
  To compare the relationship between serum AMH and ovarian response for IVF with the GnRH antagonist protocol in patients who are carriers of FSH and/or LH receptor polymorphisms with those that are not.

SECONDARY OUTCOMES:
polymorphisms in the FSH receptor (FSHR) variant N680S | 1 year
  To define the incidence of carriers of polymorphisms in the FSH receptor (FSHR) variant N680S (homozygous and heterozygous) among women undergoing ovarian stimulation for IVF.
polymorphisms in the LH receptor (LHR) variant N312S | 1 year
  To define the incidence of carriers of polymorphisms in the LH receptor (LHR) variant N312S (homozygous and heterozygous) among women undergoing ovarian stimulation for IVF.
Doses of gonadotrophin needed and polymorphisms | 1 year
  To analyse the doses of gonadotrophins needed for stimulation on each group of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Valencian Institute of Infertility, IVI RMA. Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided